CLINICAL TRIAL: NCT03886363
Title: Effectiveness of Mindfulness-Based Stress Reduction Among Danish School Teachers
Brief Title: Effectiveness of MBSR Among School Teachers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05032019
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Stress Reduction; Mental Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): MBSR according to international standards (2.5 hours group session once a week in 8 weeks; a silence retreat day; and 45-60 minutes homework six days a week). Content in accordance with MBSR curriculum.
  Interventions: Behavioral: MBSR
- Wait-list control (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: MBSR — Described previously
  Arms: MBSR

SUMMARY:
The aim is to evaluate the effectiveness of Mindfulness-Based Stress Reduction among school teachers in Danish schools on mental weii-being in the teachers and their pupils. The study is a cluster-randomised trial including 150 schools; 200 teachers; 4000 pupils from the five geographical regions in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* School teacher at a Danish school that commit to participate in a trial aiming to implement and evaluate the effectiveness of ".b" (a school-based mindfulness programme)

Exclusion Criteria:

* acute treatment-demanding clinical depression or a diagnosis of psychosis or schizophrenia
* abuse of alcohol, drugs, medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-12-18 (Estimated); Study Completion 2020-12-18 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Perceived Stress Scale
Change in resilience among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Brief Resilience Scale

SECONDARY OUTCOMES:
Change in symptoms of anxiety and depression among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Symptom Check List - 5
Change in well-being among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  WHO-5
Change in mindfulness among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Five Facet Mindfulness Questionnaire-15
Change in resting state among the school teachers | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Amsterdam Resting State Questionnaire
Change in social capital among the pupils spending >5 hours with the teachers | post MBSR (8 weeks from baseline)
  Questions about social capital
Change in strengths and difficulties among the pupils spending >5 hours with the teachers | post MBSR (8 weeks from baseline)
  Strengths and difficulties questionnaire (SDQ)
Change in well-being among the pupils spending >5 hours with the teachers | post MBSR (8 weeks from baseline)
  WHO-5

CONTACTS AND LOCATIONS:
Overall Officials: Lone Fjorback, PhD, Study Director — Aarhus University, Danish Center for Mindfulness
Locations (1):
- Danish Center for Mindfulness, Aarhus, Denmark

REFERENCES:
- [Derived] Juul L, Bonde EH, Fjorback LO. Altered self-reported resting state mediates the effects of Mindfulness-Based Stress Reduction on mental health: a longitudinal path model analysis within a community-based randomized trial with 6-months follow-up. Front Psychol. 2023 Jun 20;14:1154277. doi: 10.3389/fpsyg.2023.1154277. eCollection 2023. PMID 37408978